CLINICAL TRIAL: NCT03692442
Title: Evaluation of Efficacy and Toxicity of Nivolumab Monotherapy for Advanced Non-small Cell Lung Cancer After First-line Treatment Failure Based on Second-generation Sequencing and Liquid Chip Platform
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Guangzhou Institute of Respiratory Disease (Other)
Collaborators: GeneCast Biotechnology Co., Ltd. (Industry)
Responsible Party: Principal Investigator, ShiYue Li, Director，Guangzhou Institute of Respiratory Disease, Guangzhou Institute of Respiratory Disease
Other Study IDs: LCIO
Record Dates: First submitted 2018-09-25; First posted 2018-10-02 (Actual); Last update posted 2018-10-02 (Actual); Status verified 2018-09

CONDITIONS: Lung Cancer Non-small Cell Stage IV
Keywords: NGS; cytokine; efficacy; side effect
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- immunotherapy effective group: PD1, TMB and serum cytokines was detected before nivolumab treatment
- immunotherapy ineffective group: PD1, TMB and serum cytokines was detected before nivolumab treatment

SUMMARY:
In order to understand the efficacy and side effects of lung cancer immunotherapy, at least 30 patients with lung cancer who were treated with immunotherapy were enrolled. The second-generation sequencing technology and liquid phase factor platform were used for detection, and clinical imaging and other evaluation methods were used to explore the immunotherapy efficacy and side effects affecting lung cancer。

DETAILED DESCRIPTION:
In order to understand the efficacy and side effects of lung cancer immunotherapy, at least 30 patients with lung cancer who were treated with immunotherapy were enrolled. The second-generation sequencing technology and liquid phase factor platform were used for detection, and clinical imaging and other evaluation methods were used to explore the immunotherapy efficacy and side effects affecting lung cancer。

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be willing and able to comply with the schedule of visits, treatment protocols, laboratory tests, and other requirements of the study.
* PS > 2, lung cancer in the elderly (less than 65 years old).
* subjects' characteristics and target disease characteristics Histologically or cytologically diagnosed as NSCLC (SQ or NSQ) and with stage IIIB/IV tumors (International Association for the Study of Lung Cancer Staging Manual in Thoracic Oncology, Version 8) or multimodal therapy (radiotherapy, surgical resection) Subjects who relapsed or developed disease after radical chemoradiotherapy for locally advanced diseases.
* Prior radiotherapy or radiosurgery must have been completed at least 2 weeks prior to starting study treatmen

Exclusion Criteria:

* Women with a positive pregnancy test at enrollment or prior to administration of study medication
* Participants with a condition requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalent) or other immunosuppressive medications within 14 days of first dose of study drug
* Participants with previous malignancies are excluded unless a complete remission was achieved at least 2 years prior to study entry AND no additional therapy is required or anticipated to be required during the study period
* Participants with carcinomatous meningitis Other protocol defined inclusion/exclusion criteria could apply

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: advance lung cancer
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2018-05-01 (Actual); Primary Completion 2019-01-31 (Estimated); Study Completion 2019-03-31 (Estimated)

PRIMARY OUTCOMES:
PD-L1 expression levels | before drugs thearpy
  The positive rate of PD-L1 expression in tumor tissues was detected by immunohistochemistry
PD-1 expression levels | before drugs thearpy
  The positive rate of PD-L1 expression in tumor tissues was detected by immunohistochemistry
tumor mutation burden | before drugs thearpy
  Detection of the average number of mutations per megabyte in tumor tissues by NGS
Serum cytokine levels | before drugs thearpy
  Detect the expression level of cytokines in serum
Objective Response Rate (ORR) by irRC and RECIST 1.1 | 6 months
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Guangzhou Institute of Respiratory Disease, The First Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No